CLINICAL TRIAL: NCT05417347
Title: he Role of Full-fat Dairy Products on Body Weight Control and Metabolic Health in Adults and Children
Brief Title: Full-fat Dairy Products, Body Weight Control and Metabolic Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Vicky Drapeau, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DAIRY-2019-397
Record Dates: First submitted 2022-04-08; First posted 2022-06-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: low-fat dairy products; full-fat dairy products; weight loss and maintenance
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Masking Description: This study will be single-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-fat dairy products (Active Comparator): Consumption of low-fat dairy products (4 servings/day with 2 servings/day coming from yogurt)
  Interventions: Other: Low-fat dairy products
- Full-fat dairy products (Active Comparator): Consumption of high-fat dairy products (4 servings/day with 2 servings/day coming from yogurt)
  Interventions: Other: Full-fat dairy products
- Control (No Intervention): Will be recommended to choose low-fat dairy products and alternatives based on recommendations from the 2007 Canadian Food Guide (2 servings/day for adults and 3-4 servings/day for children)

INTERVENTIONS:
Other: Low-fat dairy products — Milk: low fat (less than 2% M.F.) Yogurt: less than 2% M.F. Cheese: less than 20% M.F.
  Arms: Low-fat dairy products
Other: Full-fat dairy products — Milk: full-fat milk Yogurt: 2% and more M.F. Cheese: Regular cheese products
  Arms: Full-fat dairy products

SUMMARY:
The aim of this research is to clarify the role of different dairy products including both full-fat and low-fat dairy in maintaining health in adults and children through its effects beyond their well-known contribution of healthy nutrients. The deleterious health consequences of obesity are recognized as a major financial burden to health care systems. Diets rich in fruits and vegetables and that also include dairy products have been suggested to play a role in the control of body weight and other aspects of health including the maintenance of healthy gut bacteria. In contrast, full-fat diets, especially those high in saturated fat, have been linked with negative health effects. Although dairy products represent an important source of saturated fat, it has been proposed that the combination of nutrients and complex food forms of the various dairy products may in fact counteract the negative effects of the fat. Thus, increased consumption of dairy products could very likely provide a partial dietary solution to improved body weight and metabolic health. Therefore, we are investigating the role of both full-fat and low-fat dairy products in their different physical forms (i.e. varying levels of fat that contribute to different textures) on appetite, food intake, control of blood sugar (glucose), body weight, cholesterol levels, and blood pressure in both children and adults. Existing dairy products (milk, cheese, and yogurt) ranging in fat content will be compared for their effects on satiety, food intake, glucose, insulin, satiety hormones, gut bacteria and other metabolic parameters linked to cardiometabolic health in normal weight children and adults, as well as in children and adults living with overweight and obesity.

DETAILED DESCRIPTION:
The overall objective is to examine the long-term effects of full-fat dairy products on appetite and body weight control, diet quality, and metabolic health in adults living with obesity (18-55 y) and in children (8-16 y). This project also aims to identify some key mechanisms (i.e. gut peptides, gut microbiota) involved in the beneficial impact of dairy products on these outcomes. This study aims to evaluate the impact of a web-based nutrition intervention integrating full-fat or low-fat dairy products into the diets of families (at least one parent with BMI >30 kg/m2) under free-living conditions, on overall dairy consumption, body weight and composition, diet quality, eating and psychobehavioural traits and cardiometabolic outcomes, in normal weight/obese adults and children. This is a randomized, controlled, single-blind study consisting of three parallel groups. Families (n=25/group) will be randomized to either an intervention promoting either 1) low-fat or 2) full-fat dairy) or 3) control group (no intervention but same follow-up) over an 8-week period. The nutrition intervention aims to increase the quantity and variety of dairy products (i.e. low and full-fat milk, yogurt and cheese) in the diet. Evaluation periods for each family will be conducted before the study (week 0 in the lab), at the end (week 9 at home) and after 3 months (week 20 at home) after the intervention. Measurements include anthropometry, fasting lipid and glycemic profiles, diet quality, eating and psychobehavioral traits and food reward/appreciation/acceptance. The proposed research will provide timely data required to support recommendations to consume low and full-fat dairy products in individuals living with obesity, particularly during weight loss and maintenance. It will also provide the basis for family interventions that have the potential to positively impact diet quality and dairy consumption.

ELIGIBILITY:
Inclusion Criteria:

Parent criteria are as follows:

* men and women between 18-55 years
* body mass index (BMI) between 30-40 kg/m2
* absence of pregnancy, breastfeeding or menopause (no menstruation)
* stable body weight (weight change <5 kg for three months prior to screening).

Family criteria are as follows:

* being a family composed of at least one parent (mother/father) and at least two children between 8 to 16 years old (families between 3 to 5 persons). Families with at least one obese parent (BMI between 30-40 kg/m2) will be recruited since children coming from these families are more at risk of developing obesity and may benefit more from dairy products
* all participants should have no allergies to dairy products or lactose intolerance and be in good general health.
* since we are recruiting adults with obesity and dairy products may positively impact several metabolic markers, those with hypertension or deteriorated blood glucose and lipid profiles and/or taking medications will also be considered.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-06-19 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Dairy consumption | 8 weeks
  # of servings of dairy

SECONDARY OUTCOMES:
Body weight (kg) | week 0, week 9, week 24
  Body weight will be measured using standard laboratory methods
Systolic and diastolic blood pressure (mmHg) | week 0, week 9, week 24
  Blood pressure will be measured using standard laboratory methods
Plasma lipids (total cholesterol, HDL and LDL cholesterol, triglycerides) | week 0, week 9, week 24
  Plasma lipids will be measured using standard laboratory methods
Gastrointestinal peptides and hormones | week 0, week 9, week 24
  The following hormones will be measured: adiponectin, amylin, leptin, ghrelin, glucose insulinotropic peptide (GIP), glucagon-like peptide (GLP-1), peptide tyrosine tyrosine (PYY), cortisol
Oral microbiota (bacterial DNA from saliva) | week 0, week 9, week 24
  Saliva samples will be collected.
Habitual food intake and diet quality | week 0, week 9, week 24
  24-h web-based dietary recalls
Eating behaviours | week 0, week 9, week 24
  Various validated questionnaires (e.g. Three-Factor Eating Questionnaire and Child Three-Factor Eating Questaionnaire) will be used to assess these traits
Physical activity | week 0, week 9, week 24
  Physical activity diary
Cravings | week 0, week 9, week 24
  All adult participants will complete the State/Trait Food Cravings Questionnaire to examine eating behaviour traits and factors which could influence appetite control and metabolic variables such as restraint behaviour and sleep deprivation. Each parent will complete the child's feeding questionnaire and the caregiver feeding style questionnaire to assess parental feeding practices.
Sleeping Habits | week 0, week 9, week 24
  Pittsburgh Sleep Quality Index Questionnaire
Resting metabolic rate | week 0, week 9, week 24
  Indirect calorimetry will be used
Binge Eating Tendencies | week 0, week 9, week 24
  All adult participants will complete the Binge Scale to examine eating behaviour traits and factors which could influence appetite control and metabolic variables such as restraint behaviour and sleep deprivation. Each parent will complete the child's feeding questionnaire and the caregiver feeding style questionnaire to assess parental feeding practices.
Cognitive restraint, disinhibition, susceptibility to hunger | week 0, week 9, week 24
  All adult participants will complete the Three Factor Eating Questionnaire to examine eating behaviour traits and factors which could influence appetite control and metabolic variables such as restraint behaviour and sleep deprivation. Each parent will complete the child's feeding questionnaire and the caregiver feeding style questionnaire to assess parental feeding practices.
Distress-related body esteem | week 0, week 9, week 24
  All adult participants will complete the Body Esteem Scale to examine eating behaviour traits and factors which could influence appetite control and metabolic variables such as restraint behaviour and sleep deprivation. Each parent will complete the child's feeding questionnaire and the caregiver feeding style questionnaire to assess parental feeding practices.
Depression symptoms | week 0, week 9, week 24
  All adult participants will complete the Beck Depression Inventory.
Anxiety symptoms | week 0, week 9, week 24
  All adult participants will complete the State-Trait Anxiety Inventory.
Stress levels | week 0, week 9, week 24
  All adult participants will complete the Perceived Stress Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Drapeau, PhD, RD, Principal Investigator — Laval University; Angelo Tremblay, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada